CLINICAL TRIAL: NCT03812341
Title: SINGLE PATIENT EXPANDED ACCESS OF A PROSPECTIVE, MULTICENTER CLINICAL TRIAL DESIGNED TO EVALUATE THE SAFETY AND PROBABLE BENEFIT OF THE KERAKLEAR NON-PENETRATING KERATOPROSTHESIS IN SUBJECTS WITH CORNEAL OPACITY WITH POOR PROGNOSIS FOR CORNEAL TRANSPLANT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-4549
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: CORNEAL OPACITY WITH POOR PROGNOSIS FOR CORNEAL TRANSPLANT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Other: Experimental — KeraKlear Non-Penetrating Keratoprosthesis The KeraKlear is a flexible non-penetrating artificial cornea designed to be implanted through small corneal incisions in subjects with corneal opacity

SUMMARY:
This is for a "Single Patient Expanded Access" of an on-going study (IRB#2017-3526). In the on-going study, the maximum number of subject will be 35 subjects (35 eyes) will be implanted with the KeraKlear device and will be followed for one year. However, this expanded access is for single patient use below is a description of patient condition and circumstances necessitating treatment:

88 year old female with 2 previous failed corneal transplants, had significant scarring and mild edema, surface well epithelialized, has potential for 10 letters of improvement in visual acuity. Patient is high risk for recurrent corneal rejection and failure and therefore would not be a candidate for standard corneal transplant. She would potentially do well with a partial thickness artificial cornea such as the KeraKlear.

DETAILED DESCRIPTION:
For this "Single Patient Expanded Access" the research procedures will be based on the Master Protocol Version #1.2 dated 18Dec2017, with one foreseen deviation. Section 7.1 Page 27 under Inclusion Criteria #1 Male or female from 22 years to 80 years of age at screening study visit. This patient is 88 years old as of the submission of this Protocol Narrative to the IRB.

Postoperatively, subject will be examined at (with window size in parentheses):

* 1 Day (+2 days)
* 1 Week (7±2 days)
* 1 Month (30±5 days)
* 2 Months (60±7 days)
* 3 Months (90±7 days)
* 4 Months (120±10 days)
* 6 Months (180±10 days)
* 9 Months (270±20 days)
* 12 Months (360±20 days)

ELIGIBILITY:
Inclusion Criteria:

* Corneal blindness where cornea transplantation is necessary but is expected to be unsuccessful due to severe limbal stem cell deficiency (LSCD) associated with aniridia or due to multiple (two or more) failed cornea transplantation surgeries and spontaneous visual improvement without surgical intervention is not expected or probable.
* Best Corrected Distance Visual Acuity (Snellen) which is equal or worse than 20/200 in the study eye (but at least light perception with projection)
* Estimated visual potential of the study eye is greater than or equal to at least two lines visual improvement of BCDVA of current vision in the study eye.

Exclusion Criteria:

* Visual Acuity of No Light Perception (NLP) in the study eye
* The patient is monocular or the non-study eye has Best Corrected Distance Visual Acuity (Snellen) of worse than 20/160 due to an ocular condition other than severe aniridic limbal stem cell deficiency or due to multiple (two or more) failed cornea transplantation surgeries.
* Suitable for standard PK with donor tissue in the study eye.
* History of severe dry eye syndrome or a Schirmer test with results of less than 3mm after 5 minutes of testing with the use of topical anesthetic in either eye.
* Active or history of an auto-immune disease (e.g. Rheumatoid Arthritis, Ocular Cicatricial Pemphigoid, Lupus, Steven's Johnson Syndrome, atopic keratoconjunctivitis, etc.).
* On medications that may affect wound healing, such as antimetabolites or other chemotherapeutic agents.
* History of posterior segment eye disease in either eye (including macular degeneration, optic neuropathy, posterior uveitis) which is expected to limit the visual improvement to less than two lines of vision.
* History of retinal surgery in the fellow eye (including retinal detachment repair, intravitreal injection etc.).
* History of retinal surgery in the study eye (including retinal detachment repair, intravitreal injection, etc.) unless the vision is at least light perception with projection in four field quadrants and the macula is attached (if there is no view of the retina, an ultrasound must show the macula is attached).
* History of uncontrolled glaucoma in either eye (IOP has been measured above 25 mmHg at any time in the last 6 months).
* Current use of beta blocker eye drops (e.g. timolol, levobunolol, etc.).
* Vertical cup-to-disc (C:D) ratio greater than or equal to 0.8 in either eye (if able to visible through corneal opacity). If not visible, patient is not to be excluded.
* Limited visual potential (patient does not have the ability to improve a minimum of two lines of vision of BCDVA by history).
* History of amblyopia in the study eye limiting visual potential.
* If the patient has had a corneal transplant, corneal transplantation surgery was performed less than 2 years ago.
* Anticipated need for surgery on the study eye during the course of the study (including cataract surgery).
* Aphakia in the study eye.
* Active ocular infection in either eye.
* Hypotony in the study eye (IOP < 6mmHg).
* History of herpetic ocular infection in the study eye.
* Corneal thickness less than 400 microns in any region of the pachymetry map.
* Inability to protect the operated eye from trauma.
* Females who are pregnant, lactating, or unwilling to use adequate birth control for t the duration of the study.
* Patient is currently taking Sumatriptan (Imitrex) and unable to discontinue during the study.

For this "Single Patient Expanded Access" the research procedures will be based on the Master Protocol Version #1.2 dated 18Dec2017, with one foreseen deviation. Section 7.1 Page 27 under Inclusion Criteria #1 Male or female from 22 years to 80 years of age at screening study visit. This patient is 88 years old.

-

Ages: 88 Years to 88 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — 88 year old female.
Enrollment: 0 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
1.Improvement in BCDVA compared to baseline [ Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 6, Month 9 and Month 12 ] | 1 year
  Best Corrected Distance Visual Acuity (BCDVA) will be measured in the study eye. An ETDRS visual acuity chart will be used to measure BCDVA at baseline, Month 1, Month 2, Month 3, Month 4, Month 6, Month 9, and Month 12.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No